CLINICAL TRIAL: NCT00690326
Title: Behavioral Change Communication to Promote Physical Activity Among Females With Type 2 Diabetes Mellitus Attending Diabetic Clinic.
Brief Title: Behavioral Change Communication (BCC) to Promote Physical Activity Among Females With Type 2 Diabetes Mellitus Attending Diabetic Clinic
Acronym: BCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thiruvananthapuram Medical College (Other)
Responsible Party: Dr. Rose Dvy.C, Assistant professor Dept. Physiology,Thiruvananthapuram Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Physical activity RCT
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: physical activity; Diabetes mellitus; Behavioral change communication; Household physical activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): treatment type: behavioral(lifestyle counseling)
  treatment name: behavioral change communication to promote physical activity
  Interventions: Behavioral: Behavioral change communication to promote physical activity
- B (Placebo Comparator): Arm B given placebo comparator ie pamphlets
  Interventions: Behavioral: Behavioral change communication to promote physical activity

INTERVENTIONS:
Behavioral: Behavioral change communication to promote physical activity — treatment type: behavioral (lifestyle counseling)
  treatment name: behavioral change communication to promote physical activity
  Arms: A
Behavioral: Behavioral change communication to promote physical activity — Arm B given placebo comparator ie pamphlet
  Audiovisual module Physical activity frequency questionnaire
  Arms: B

SUMMARY:
Type 2DM is present in the populations of almost all the countries in the world and is a significant disease burden in most countries .Evidences suggest that population in India develop Type 2 DM at an increasing rate as they reject their traditional life styles.

Awareness and knowledge regarding Diabetes and role of physical inactivity in producing complications is still grossly inadequate( Mohan. D, Raj.D Awareness and knowledge of Diabetes in Chennai.The Chennai urban Rural Epidemiology study(CURES-9)J Assoc. Physicians India 2005 April;53:283-7).Exercise is a low cost , non pharmacological intervention that has been shown to be effective in metabolic control. Exercise is still vastly under-utilized in the management of Type 2 DM.

Most proximal behavioral cause of insulin resistance is physical inactivity.(Michael J. LaMonte, Steven N. Blair et al.( Physical activity and Diabetes prevention J Appl Physiol. 99: 1205-1213,2005)

This study was designed to promote physical activity among type 2 DM female subjects aged 35-65 yrs attending Diabetic clinic of a tertiary care hospital in Kerala.

DETAILED DESCRIPTION:
The BCC model consisted of 1.an audio visual module imparting knowledge about DM, its complications, advantages of PA in Diabetes control, how to include more PA in routine life style 2. pamphlets.All these were standardised. Physical activity was measured using international physical activity questionnaire validated(responsiveness& reliability) for our cultural activity.IPAQ covers four domains of physical activity: work-related,transportation, housework/gardening and leisure-time activity. PA data from the questionnaire were transformed into energy expenditure estimates as MET using published values. To calculate the weekly physical activity (MET-h /week), the number of hours dedicated to each activity class was multiplied by the specific MET score for that activity.

follow up once in a month (4 times) measure incremental physical activity and reinforcement in each visit. Students t test was used to compare the experimental and control groups with respect to the incremental physical activity measured in calorie expenditure. It was found that the incremental physical activity(final-basal) measured in METS is significantly higher in intervention group.

ELIGIBILITY:
Inclusion Criteria:

* females 30to 65yrs. with type-2 Diabetes Mellitus.
* Attending Diabetic clinic at a tertiary level hospital(medical college Thiruvananthapuram)
* on oral hypoglycemics

Exclusion Criteria:

* only one patient from one family
* H/o myocardial infarction
* nephropathy
* autonomic neuropathy
* severe limiting osteo arthritis
* pregnancy
* Mental incompetence

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-05; Primary Completion 2006-07 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
incremental physical activity | at the end of 4 months-October

SECONDARY OUTCOMES:
glycosylated hemoglobin | At the end of 4 months -October

CONTACTS AND LOCATIONS:
Overall Officials: Rose D Chakola, MD MPhil, Principal Investigator — CERTC-Clinical epidemiology research&training centre,Trivandrum medical college
Locations (1):
- Diabetic clinic,Thiruvananthapuram medical college hospital, Thiruvananthapuram, Kerala, India